CLINICAL TRIAL: NCT07159334
Title: Role of Topical Application of Lignocaine Versus 0.2% Glyceryl Trinitrate (GTN) Ointment as a Postoperative Local Analgesic in Hemorrhoidectomy in Terms of Pain Score,Wound Healing Time and Patient Satisfaction Level
Brief Title: "Lignocaine vs GTN Ointment for Postoperative Pain After Hemorrhoidectomy")
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahmad Rauf
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hemorrhoid; Postoperative Pain
Keywords: Hemorrhoidectomy; Lignocaine ointment; Glyceryl Trinitrate ointment; Anal pain
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: "Participants will be randomized into two parallel groups: one receiving topical lignocaine ointment and the other receiving topical glyceryl trinitrate ointment for postoperative pain management after hemorrhoidectomy."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1.Lignocaine Ointment Group (Experimental): Participants will receive topical lignocaine ointment applied to the anal wound post-hemorrhoidectomy for pain control.
  Interventions: Drug: Lignocaine Ointment; Drug: Glyceryl Trinitrate Ointment 0.2%
- Glyceryl Trinitrate Ointment Group (Experimental): Participants will receive topical 0.2% glyceryl trinitrate ointment applied to the anal wound post-hemorrhoidectomy for pain control.
  Interventions: Drug: Lignocaine Ointment; Drug: Glyceryl Trinitrate Ointment 0.2%

INTERVENTIONS:
Drug: Lignocaine Ointment — Applied to the anal wound three time daily after hemorrhoidectomy.
Drug: Glyceryl Trinitrate Ointment 0.2% — Applied to the anal wound three time daily after hemorrhoidectomy.

SUMMARY:
This study is being conducted at the Department of General Surgery, King Edward Medical University, Lahore, Pakistan. The purpose of the trial is to compare the effectiveness of topical Lignocaine ointment versus topical Glyceryl Trinitrate (GTN) ointment in reducing postoperative pain following hemorrhoidectomy.

Patients undergoing hemorrhoidectomy will be randomly assigned to receive either Lignocaine ointment or GTN ointment applied locally after surgery. Pain relief will be assessed using a visual analog scale (VAS) at regular intervals during the postoperative period. The study aims to determine which ointment provides better pain control and improves patient comfort during recovery.

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of lignocaine versus 0.2% glyceryl trinitrate (GTN) ointment as postoperative analgesics in patients who have undergone hemorrhoidectomy.

Background

Hemorrhoids are swollen veins in the anal region, commonly treated through Milligan-Morgan hemorrhoidectomy. Postoperative pain is a major concern, affecting mobility and delaying recovery.

Various treatments have been explored to alleviate post-hemorrhoidectomy pain, including anal dilatation, NSAIDs, opioids, and topical treatments like nifedipine, botulinum toxin, lignocaine, and GTN ointment.

Both GTN and lignocaine have been shown to reduce pain, but the most effective and safe option is still unclear.

Study Objective

To compare the outcomes of lignocaine versus 0.2% GTN ointment in reducing pain and promoting wound healing in post-hemorrhoidectomy patients.

Hypothesis

There is a difference in the pain relief and wound healing outcomes between lignocaine and GTN ointment in hemorrhoidectomy patients.

Study Design

Randomized clinical trial conducted at the Department of Surgery, Mayo Hospital, Lahore.

Duration: 3-6 months after synopsis approval.

Sample Size: 64 patients (32 in each group).

Inclusion Criteria: Age 18-60, both genders, Grade III/IV hemorrhoids, ASA grades I & II.

Exclusion Criteria: Allergies to lignocaine or GTN, pregnancy, concomitant perianal pathology, cardiovascular issues, use of nitrates or calcium channel blockers.

Methods

Participants will undergo hemorrhoidectomy under spinal anesthesia/saddle block/general anesthesia.

Group A will receive lignocaine cream, and Group B will receive 0.2% GTN ointment post-operatively (applied 3 times daily).

Both groups will receive standard postoperative care (sitz baths, stool softeners, and paracetamol for pain).

Outcome Measures:

Pain Score using Visual Analogue Scale (VAS) at various time points (6, 12, 24, 48, 72 hours; 7, 14, 21, and 28 days post-surgery).

Time to complete wound healing (measured in days).

Level of patient satisfaction after 6 weeks using a 5-point Likert scale.

Data Analysis

Data will be analyzed using SPSS. Descriptive statistics for quantitative variables (e.g., age, pain scores) and qualitative variables (e.g., gender, patient satisfaction).

Independent t-tests will be used to compare outcomes between groups. A p-value < 0.05 will be considered statistically significant.

Patient Follow-Up

Patients will be followed for 6 weeks post-surgery to monitor pain levels, wound healing, and satisfaction.

Conclusion

This trial aims to determine which topical analgesic-lignocaine or GTN ointment-is more effective for postoperative pain management and wound healing in hemorrhoidectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 60 years
* Both genders
* Grade III and IV hemorrhoids diagnosed on the basis of history and clinical examination by consultant Surgeon.(Grade III Hemorrhoid manually reduced by patient with finger and Grade IV is prolapsed)
* ASA (American society of Anesthesia) grades I, and II

Exclusion Criteria:

* Previously reported allergy or reaction to lignocaine and GTN
* Pregnancy or lactation
* Concomitant perianal pathology warranting surgery
* Cardiovascular disease
* Patient taking Nitrates or Calcium channel blocker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-08-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | Up to 1 month postoperatively.
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain severity.
Wound Healing Time | Up to 1 month postoperatively.
  Defined as the number of days from the date of surgery until complete wound healing (full epithelialization with no discharge or open area). Shorter duration indicates a better outcome.

SECONDARY OUTCOMES:
patient Satisfaction Level | 6 weeks postoperatively
  Overall satisfaction with postoperative care and treatment, assessed using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied). Higher scores indicate greater satisfaction.
Time to Request of First Analgesic Dose | Within 24 hours postoperatively
  Time (in minutes/hours) from end of surgery to first request for analgesia. Shorter time indicates earlier need for pain control.
Amount of Analgesia Administered in First 24 Hours | 0-24 hours postoperatively
  Total rescue analgesic dose administered in first 24 hours, recorded in mg (converted to morphine-equivalent dose if applicable). Lower values indicate better pain control.
Incidence of Wound Secretion | 1 month postoperatively
  Presence of wound secretion (yes/no) as noted on clinical examination.
Incidence of Itching | 1 month postoperatively
  Patient-reported pruritus at wound site (yes/no)
Incidence of Postoperative Bleeding | 1 month postoperatively
  Occurrence of wound bleeding postoperatively (yes/no).
Incidence and Severity of Headache | 1 month postoperatively
  Patient-reported headache severity measured using a Numerical Rating Scale (0 = no headache, 10 = worst imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz Ahmad Rauf, Principal Investigator — King Edward Medical University/Mayo hospital Lahore
Locations (1):
- King Edward Medical uUniveristy Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT07159334/Prot_SAP_000.pdf